CLINICAL TRIAL: NCT03205124
Title: The Effect of Pre-operative And/or Post-operative Electrical Stimulation on Enhancing Regeneration of Peripheral Sensory Nerve Regeneration in Human Hand, a Double Blind Randomized Controlled Study.
Brief Title: The Effect of Pre-operative Electrical Stimulation on Peripheral Nerve Regeneration.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UAlberta Pre-Conditioning
Record Dates: First submitted 2017-06-25; First posted 2017-07-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Nerve Injuries; Sensory Deficit; Digital Nerve Lesion
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Three arm randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-operative stimulation (Experimental): Patients randomized to this group will receive 1 hour of continuous electrical stimulation three days prior to scheduled surgical date. The frequency will be fixed at 20Hz and the voltage and duration of electrical pulses will be sequentially increased to the maximum tolerable limit. As the nerve becomes accustomed to the sensation of the stimulation, the voltage is increased to the next tolerable threshold and this is repeated throughout the one-hour period. Once the stimulation is complete, the stimulator is detached and the patient is informed of the surgical date. The wires are taken out at the conclusion of the pre-operative appointment. These patients will have fine gauge wires for post-operative sham stimulation implanted at the time of surgery. In the post-operative recovery room the stimulator is attached to their wires. However, the voltage will only be increased to a level they are able to sense.
  Interventions: Procedure: Electrical Stimulation
- Sham stimulation (Sham Comparator): These patients will have the stimulator attached to their wires 3 days prior to scheduled surgical date and postoperatively as were in the previous groups. However, the voltage will only be increased to a level they are able to sense. The stimulator was then be turned off without the patients' knowledge. All connections are left in place for anhour duration. These patients will similarly have their wires removed after the conclusion of their pre-operative appointment and at the first post-operative follow-up within 1 week of surgery.
  Interventions: Procedure: Sham Stimulation
- Pre and Post-operative stimulation (Experimental): Patients randomized to this group will receive 1 hour of continuous electrical stimulation three days prior to scheduled surgical date and then again immediately post operatively. The frequency will be fixed at 20Hz and the voltage and duration of electrical pulses will be sequentially increased to the maximum tolerable limit. As the nerve becomes accustomed to the sensation of the stimulation, the voltage is increased to the next tolerable threshold and this is repeated throughout the one-hour period. Patients randomized to this group will also receive 1 hour of continuous electrical stimulation post-operatively. These patients will have fine gauge wires for post-operative stimulation implanted at the time of surgery. In the post-operative recovery room the stimulator is attached to their wires. The frequency will be fixed at 20Hz and the voltage and duration of electrical pulses will be sequentially increased to the maximum tolerable limit for one hour.
  Interventions: Procedure: Electrical Stimulation

INTERVENTIONS:
Procedure: Electrical Stimulation — The experimental treatment involves implantation of 2 sterilized fine-gauge Teflon coated wires percutaneously. The ends of the wire are stripped for conductivity. Electrical stimulation is given at a fixed continuous frequency of 20Hz. The stimulus intensity is the maximum tolerable limit. The wires are then taped to the skin with surgical wound tape at a location away from the wound for strain relief. To ensure sterility, care is taken to dress the sutured wound and hand, as well apply the splint.
  The wires are removed either immediately at the conclusion of the pre-operative appointment and immediately after surgery or at the first surgical follow-up with dressing change, within one week of surgery.
  Arms: Pre and Post-operative stimulation; Pre-operative stimulation
Procedure: Sham Stimulation — The experimental treatment involves implantation of 2 sterilized fine-gauge Teflon coated wires percutaneously. The ends of the wire are stripped for conductivity. Electrical stimulation is begun until the patient senses the stimulation, then the stimulation is discontinued.The wires are then taped to the skin with surgical wound tape at a location away from the wound for strain relief. To ensure sterility, care is taken to dress the sutured wound and hand, as well apply the splint.
  The wires are removed either immediately at the conclusion of the pre-operative appointment and immediately after surgery or at the first surgical follow-up with dressing change, within one week of surgery.
  Arms: Sham stimulation

SUMMARY:
Traumatic injury to the peripheral nerves is most common in the young population with high associated costs to the patient, as well as to society. These range from acute healthcare cost to loss of productivity and rehabilitation. Despite major efforts in improving surgical technique, functional outcome has not significantly improved in the past thirty years. Irreversible denervation, atrophy of target muscles, and deranged sensation secondary to slow or aberrant axonal outgrowth remains a significant challenge. Although pre-operative conditioning of the injured peripheral nerve with electrical stimulation has shown promise in animal studies, it has not been tested in humans.

In animal studies, pre-operative conditioning with electrical stimulation (ES) of the injured peripheral nerves promoted peripheral nerve regeneration in both sensory and motor fibres. We propose to conduct a clinical trial comparing 3 different treatments of complete digital nerve laceration before and after surgical repair. Participants will be randomized to one of three treatment arms: i) pre and post operative electrical stimulation, ii) pre-operative electrical stimulation alone , or iii) control group that receives sham pre and post-operative electrical stimulation. We will evaluate the effect of pre-operative electrical stimulation on axonal regeneration, as well as determine whether there is an additive effect of pre and post-operative electrical stimulation on sensory nerve axonal regeneration.

DETAILED DESCRIPTION:
Purpose:

The purpose of this research study is to determine the effect of pre-operative electrical stimulation (ES) on sensory nerve regeneration in the digital nerves that have been traumatically transected and subsequently surgically repaired.

Hypothesis:

Based on previous animal and human research, we hypothesize that pre-operative ES will result in significant improvement of sensory nerve regeneration in the hand compared to surgery alone after a traumatic digital nerve laceration. Additionally, we hypothesize that pre-operative along with post-operative ES will have an additive effect on sensory nerve regeneration compared to pre-operative ES and surgery alone.

Justification:

Traumatic injury to the peripheral nerves is most common in the young population; therefore resulting disability incurs a significant cost to the patient, as well as to society, from loss of productivity and healthcare dollars spent on rehabilitation. Despite major efforts in improving surgical technique, functional outcome has not significantly changed in the past thirty years. Irreversible denervation, atrophy of target muscles, and deranged sensation secondary to slow or aberrant axonal outgrowth remains a significant challenge. Currently the application of post-operative electrical stimulation is being used to promoted axonal regeneration to good effect. However, pre-operative conditioning of the injured peripheral nerve, with electrical stimulation, has not been investigated in the human population.

Pre-operative conditioning with electrical stimulation (ES) of the injured peripheral nerves demonstrates particular promise. The mechanism of action of conditioning lesions consists of up regulation of regenerative associated genes and the cAMP and JAK/STAT pathways. Data from animal models, examining the effect of pre-operative electrical stimulation of peripheral nerves, demonstrate that this technique promotes peripheral nerve axonal regeneration. Senger et al have demonstrated that electrical stimulation produced axonal regeneration that is equivalent to the traditional pre-conditioning crush lesion. Thus, electrical stimulation has been proven as a viable method of pre-conditioning peripheral nerves, in order to promote upregulate axonal regeneration prior to primary coaptation of the nerve. Senger et al have also investigated the mechanism of action of this improved axonal regeneration in animals pre-conditioned with electrical stimulation and have found upregulation of regenerative associated genes.

The effect of post-operative electrical stimulation on surgically repaired peripheral nerves is well detailed in the literature. Thus it may be synergistic to combine pre and post-operative electrical stimulation. Previously animal work has been translated into patients with digital nerve transection and repair, and carpal tunnel syndrome. Wong et al demonstrated those patients who underwent complete digital nerve transection, surgical repair, and postoperative 1 hour of 20Hz continuous ES showed consistently greater improvements in all sensory modalities by 5 to 6 months postoperatively compared to the controls. Gordon et al demonstrated brief post-surgical ES resulted in robust motor reinnervation to the thenar muscles by 3 months whereas it took more than a year in the control patients.

Nix and Hopf demonstrated that low frequency ES of the crushed motor nerve to the soleus in rabbits accelerated improvement in muscle force production by 2 weeks compared to controls. Pocket and Gavin using the rat model showed that the toe-spray reflex in crushed sciatic nerves recovered significantly faster with low frequency and low intensity ES. Al-Majed et al showed that one hour of low frequency 20Hz ES of transected and repaired rat femoral nerves accelerated the slow-staggered regeneration growing across the repair site as well as enhanced preferential motor reinnervation. Even when the ES was delayed by up to 2 weeks post-rat femoral nerve repair, the enhancing effects were still persevered. In a companion study of the same year, those investigators showed that ES upregulated brain-derived neurotrophic factor and its receptor trkB within the first 2 days after surgery. Brushart et al showed that brief low frequency ES improves the specificity of reinnervation. Geremia et al performed a pivotal study showing an increase in axonal regeneration in sensory neurons if the period of post-surgical ES was no more than 1 hr. The effect was blunted if the stimulation period was any longer.

To date, no studies have been done to look at the effect of pre-operative conditioning on sensory reinnervation of human peripheral nerves with ES. Given the promising nature of the animal data from Senger et al, and the well documented effectiveness of post-operative electrical stimulation of surgically repaired peripheral nerves, we designed this study to evaluate the effects of pre-operative conditioning with ES, as well as pre-operative and post-operative ES on digital nerve sensory recovery post transection and repair.

Objectives:

The objectives of this study are two-fold. To determine the effect of pre-operative ES alone, as well as combined with post-operative ES on digital nerve regeneration of sensation, post-transection and surgical repair, when compared to control patients with surgery alone.

Research Method/Procedures:

Design:

This is a double-blinded randomized placebo controlled trial that tests the effect of ES on sensory (digital) nerve recovery in the human hand. Patients will be recruited in the hand trauma (Plastic Surgery) clinics across Edmonton. Once consented for the research study, the subject will undergo a battery of tests (Semmes-Weinstein Monofilament Test, 2-point discrimination, quantitative sensory testing for cold, warm and heat pain thresholds, as well as the Disability of the Arm, Shoulder and Hand [DASH] questionnaire) preoperatively to determine their baseline deficit prior to surgery.

Surgery:

All surgeons and intraoperative staff will be blinded from the experimental treatment. All procedure is the same for every patient in the operating suite. Patients will receive the standard-of-care surgical repair of their digital nerve with microscopic magnification and using fine-gauge sutures. Every patient will have 2 fine-gauge Teflon insulated wires (sterilized at the hospital where the surgery is done) inserted proximal to the nerve injury site, away from the suture site, 3 days pre-operatively and immediately post operatively. Those wires will be attached to the electrical stimulator that activates the nerve and send action potentials towards the cell body. For that reason, the patient must not receive local anesthetic because that would block the sodium channels, abolishing action potential propagation and nullify the effects of electrical stimulation.

Post-operative Recovery:

Patients will be assessed for baseline characteristics three days prior to the scheduled surgical date,l fine-gauge wires will be implanted percutaneous proximal to the presumed nerve injury site, these wires will be attached to an electrical stimulator (model SD9, Grass Instruments, Providence, RI, USA). At that point, the personnel directly connected to the study will leave the room. A research assistant who is not otherwise connected to the study will take over. An opaque envelope that contains a computed generated randomization code will be opened to determine the patient treatment group.

Treatment group A: Pre-operative stimulation with sham post-operative stimulation

Patients randomized to this group will receive 1 hour of continuous electrical stimulation three days prior to scheduled surgical date. The frequency will be fixed at 20Hz and the voltage and duration of electrical pulses will be sequentially increased to the maximum tolerable limit. As the nerve becomes accustomed to the sensation of the stimulation, the voltage is increased to the next tolerable threshold and this is repeated throughout the one-hour period. Once the stimulation is complete, the stimulator is detached and the patient is informed of the surgical date. The wires are taken out at the conclusion of the pre-operative appointment. These patients will have fine gauge wires for post-operative sham stimulation implanted at the time of surgery. In the post-operative recovery room the stimulator is attached to their wires. However, the voltage will only be increased to a level they are able to sense. The stimulator was then be turned off without the patients' knowledge. All connections are left in place. These patients will have their wires removed at the first follow-up within 1 week.

Treatment group B: Pre-operative and post-operative stimulation:

Patients randomized to this group will receive 1 hour of continuous electrical stimulation three days prior to scheduled surgical date and then again immediately post operatively. The frequency will be fixed at 20Hz and the voltage and duration of electrical pulses will be sequentially increased to the maximum tolerable limit. As the nerve becomes accustomed to the sensation of the stimulation, the voltage is increased to the next tolerable threshold and this is repeated throughout the one-hour period. Once the stimulation is complete, the stimulator is detached and the patient is informed of the surgical date. The wires are taken out at the conclusion of the pre-operative appointment. Patients randomized to this group will also receive 1 hour of continuous electrical stimulation post-operatively. These patients will have fine gauge wires for post-operative stimulation implanted at the time of surgery. In the post-operative recovery room the stimulator is attached to their wires. The frequency will be fixed at 20Hz and the voltage and duration of electrical pulses will be sequentially increased to the maximum tolerable limit. As the nerve becomes accustomed to the sensation of the stimulation, the voltage is increased to the next tolerable threshold and this is repeated throughout the one hour period. Once the stimulation is complete, the stimulator is detached and the patient is informed of the next follow-up. The wires are taken out at the first follow-up within a week with the first dressing and splint change

Sham-Placebo Control Group

These patients will have the stimulator attached to their wires 3 days prior to scheduled surgical date and postoperatively as were in the previous groups. However, the voltage will only be increased to a level they are able to sense. The stimulator was then be turned off without the patients' knowledge. All connections are left in place for a hour duration. These patients will similarly have their wires removed after the conclusion of their pre-operative appointment and at the first post-operative follow-up within 1 week of surgery.

Post-operative Follow-up:

All patients will have a one week post-operative visit, and then subsequently be followed monthly where the previously mentioned sensory nerve assessment tests as well as sensory nerve conduction studies and the Canadian Occupational Performance Measure will be done. There are a total of six monthly visits, each visit will take about 1.5h.

Sample size calculation

Based on a pivotal paper by Geremia et al; in the rat the difference in the number of regenerated sensory axons following 1h ES was 397+/-321 (SD) compared to the controls. With the type I error set at 0.05 and the type II error at 0.80, a sample size of 20 would be needed in the treatment group and the same number in the control group. To account for 10% of potential patients loss to follow-up we aim to recruit a total of 66 patients. An interim analysis will be done by the data monitoring team once the first 10 patients have completed their 6 month follow-up.

Plan for data analysis:

Per protocol analysis will be completed. All results will be reported as mean + standard deviation. Student t test and Fischer exact test will be preformed to determine demographic differences between treatment groups. Differences in sensory testing results will be evaluated via chi square testing. ANOVA will be used to determine reproducibility of testing by comparing outcomes to the contralateral hand. ANOVA variance analysis will also be preformed on all post treatment time points to determine whether the treatments differ over time. A 5% (alpha) level will be considered a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65
* with a traumatic complete transection of one or more digital nerve(s) in the hand
* and receive surgery within 2 weeks of injury.

Exclusion Criteria:

* Age <18y and >65y,
* Uncontrolled diabetes (HbA1C>8%),
* Cognitively impaired,
* Non-English speaking,
* Medically unfit for general anesthetic or personally refuse GA,
* Incomplete partial nerve lacerations,
* Crush injury,
* Concomitant bone injury in the same digit of nerve injury,
* Large nerve gap requiring graft, conduit or extreme joint flexion,
* Injury>14days prior to surgical repair,
* Patients unable to comply with 6 month follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Sensory nerve conduction studies | Change from baseline to 6 months
  An electromyography technique used to analyze sensory nerve recovery of the digital nerve.

SECONDARY OUTCOMES:
Semmes-Weinstein Monofilaments | Baseline, 1,2,3,4,5,6 months
  Measurement of pressure sensitivity
Two Point Discrimination Disk | Baseline, 1,2,3,4,5,6 months
  Measurement of spatial determination
CASE (Computer assisted Sensory Examination) | Baseline, 1,2,3,4,5,6 months
  Quantative sensory testing
Cold temperature detection threshold | Baseline, 1,2,3,4,5,6 months
DASH questionnaire | Baseline, 1,2,3,4,5,6 months
  Validated questionnaire for functionality in digital nerve injury
Vibration Threshold Testing | Baseline, 1,2,3,4,5,6 months

CONTACTS AND LOCATIONS:
Overall Officials: K Ming Chan, MB ChB, Principal Investigator — University of Alberta; Julie Beveridge, MD, Study Director — University of Alberta
Locations (2):
- Canada (2):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Salegio EA, Pollard AN, Smith M, Zhou XF. Macrophage presence is essential for the regeneration of ascending afferent fibres following a conditioning sciatic nerve lesion in adult rats. BMC Neurosci. 2011 Jan 20;12:11. doi: 10.1186/1471-2202-12-11. PMID 21251261
- [Background] Al-Majed AA, Brushart TM, Gordon T. Electrical stimulation accelerates and increases expression of BDNF and trkB mRNA in regenerating rat femoral motoneurons. Eur J Neurosci. 2000 Dec;12(12):4381-90. PMID 11122348
- [Background] Al-Majed AA, Neumann CM, Brushart TM, Gordon T. Brief electrical stimulation promotes the speed and accuracy of motor axonal regeneration. J Neurosci. 2000 Apr 1;20(7):2602-8. doi: 10.1523/JNEUROSCI.20-07-02602.2000. PMID 10729340
- [Background] Brushart TM, Jari R, Verge V, Rohde C, Gordon T. Electrical stimulation restores the specificity of sensory axon regeneration. Exp Neurol. 2005 Jul;194(1):221-9. doi: 10.1016/j.expneurol.2005.02.007. PMID 15899259
- [Background] Chan KM, Curran MW, Gordon T. The use of brief post-surgical low frequency electrical stimulation to enhance nerve regeneration in clinical practice. J Physiol. 2016 Jul 1;594(13):3553-9. doi: 10.1113/JP270892. Epub 2016 Mar 24. PMID 26864594
- [Background] Elzinga K, Tyreman N, Ladak A, Savaryn B, Olson J, Gordon T. Brief electrical stimulation improves nerve regeneration after delayed repair in Sprague Dawley rats. Exp Neurol. 2015 Jul;269:142-53. doi: 10.1016/j.expneurol.2015.03.022. Epub 2015 Apr 2. PMID 25842267
- [Background] Geremia NM, Gordon T, Brushart TM, Al-Majed AA, Verge VM. Electrical stimulation promotes sensory neuron regeneration and growth-associated gene expression. Exp Neurol. 2007 Jun;205(2):347-59. doi: 10.1016/j.expneurol.2007.01.040. Epub 2007 Feb 21. PMID 17428474
- [Background] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Background] Lundborg G. A 25-year perspective of peripheral nerve surgery: evolving neuroscientific concepts and clinical significance. J Hand Surg Am. 2000 May;25(3):391-414. doi: 10.1053/jhsu.2000.4165. PMID 10811744
- [Background] Nix WA, Hopf HC. Electrical stimulation of regenerating nerve and its effect on motor recovery. Brain Res. 1983 Aug 1;272(1):21-5. doi: 10.1016/0006-8993(83)90360-8. PMID 6616196
- [Background] Pockett S, Gavin RM. Acceleration of peripheral nerve regeneration after crush injury in rat. Neurosci Lett. 1985 Aug 30;59(2):221-4. doi: 10.1016/0304-3940(85)90203-4. PMID 3877256
- [Background] Udina E, Furey M, Busch S, Silver J, Gordon T, Fouad K. Electrical stimulation of intact peripheral sensory axons in rats promotes outgrowth of their central projections. Exp Neurol. 2008 Mar;210(1):238-47. doi: 10.1016/j.expneurol.2007.11.007. Epub 2007 Nov 22. PMID 18164293
- [Background] Wong JN, Olson JL, Morhart MJ, Chan KM. Electrical stimulation enhances sensory recovery: a randomized controlled trial. Ann Neurol. 2015 Jun;77(6):996-1006. doi: 10.1002/ana.24397. Epub 2015 May 4. PMID 25727139
- [Background] Blesch A, Lu P, Tsukada S, Alto LT, Roet K, Coppola G, Geschwind D, Tuszynski MH. Conditioning lesions before or after spinal cord injury recruit broad genetic mechanisms that sustain axonal regeneration: superiority to camp-mediated effects. Exp Neurol. 2012 May;235(1):162-73. doi: 10.1016/j.expneurol.2011.12.037. Epub 2011 Dec 29. PMID 22227059
- [Background] Moalem-Taylor G, Li M, Allbutt HN, Wu A, Tracey DJ. A preconditioning nerve lesion inhibits mechanical pain hypersensitivity following subsequent neuropathic injury. Mol Pain. 2011 Jan 5;7:1. doi: 10.1186/1744-8069-7-1. PMID 21205324